CLINICAL TRIAL: NCT00650949
Title: A Phase Ib/II Study of CYT997 in Combination With Carboplatin in Relapsed Glioblastoma Multiforme
Brief Title: Efficacy Study of CYT997 in Combination With Carboplatin in Glioblastoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Strategic
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCL08001
Record Dates: First submitted 2008-03-27; First posted 2008-04-02 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma multiforme; Glioma; Phase Ib/II; CYT997
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — CYT997; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CYT997 (Experimental)
  Interventions: Drug: CYT997; Drug: Carboplatin

INTERVENTIONS:
Drug: CYT997 — Escalating doses (100mg/m^2 to 150mg/m^2), 24-hour intravenous infusion on Day 2 of a 21-day cycle (Phase Ib component). Dose selected in Phase Ib component to be used for Phase II component.
Drug: Carboplatin — Intravenous infusion over 1 hour at area under the concentration-time curve (AUC)=5 on Day 1 of a 21-day cycle

SUMMARY:
This study seeks to (i) determine the safe dose of CYT997 when given in combination with carboplatin in patients with relapsed glioblastoma multiforme (glioma) and (ii) to determine whether the combination of CYT997 with carboplatin is a useful treatment for glioma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-confirmed glioblastoma multiforme that has progressed after initial surgery, radiation therapy and temozolomide chemotherapy.
* Measurable tumour must be present on gadolinium-enhanced MRI
* At least 3 months must have elapsed from completing radiation to minimize the possibility of pseudo-progression.
* At least 4 weeks since prior chemotherapy (6 weeks if the last regimen included bischloroethylnitrosourea (BCNU) or Chloroethyl-Cyclohexyl-NitrosoUrea (CCNU)).
* Age ≥ 18 years.
* If patients are taking steroids, the dose must be stable for = 7 days.
* Eastern Cooperative Oncology Group (ECOG) performance status = 2.
* Life expectancy of greater than 2 months.
* Patients must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count = 1.5 × 109/L
  * Platelet count = 100 × 109/L
  * Total bilirubin within normal limits
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 5 × upper limit of normal (ULN)
  * Creatinine within normal limits OR creatinine clearance = 60 mL/min/1.73 m2 for patients with creatinine levels above normal
  * Normal left ventricular ejection fraction on a gated blood pool scan or echocardiogram
* Must agree to use adequate contraceptive measures if indicated
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have received any other investigational agent in the preceding four weeks prior to commencing therapy in this study.
* Patients who have been previously treated with carboplatin.
* Patients who have been previously treated with bevacizumab or other anti-angiogenesis or vascular-disrupting agents
* Patients who are receiving enzyme-inducing anticonvulsant drugs (EIACD) such as phenytoin or carbamazepine.
* Patients with a history of allergic reactions attributed to compounds of similar chemical composition to CYT997 or other agents used in the study.
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or lactating women.
* Patients with immune deficiency, including HIV-positive patients.
* Patients with uncontrolled diarrhoea despite optimal medication and those with any history of acute gastrointestinal bleeding.
* Patients who are unable or unwilling to undergo MRI scanning
* Patients with the following conditions/treatments will be excluded:

  * Myocardial infarction (MI) or stroke within 6 months
  * History of stroke or transient ischemic attacks (TIAs)
  * Unstable angina pectoris or acute ischemic changes on ECG
  * History of diabetic retinopathy
  * Symptomatic peripheral arterial disease o Major surgery in the last 4 weeks
  * Evidence of intra-tumoural haemorrhage on imaging, except for stable grade-1 post-operative haemorrhage.
  * Current therapeutic anti-coagulation with warfarin or a heparin (excludes lowdose prophylactic heparin).
  * Uncontrolled hypertension
  * The need for any anti-arrhythmic drugs
* Presence of luminal stenosis of 50% or more in any of the extracranial or intracranial arteries supplying the brain, as measured by magnetic resonance angiography (MRA) at baseline.
* Patients with a baseline prolongation of the QTc interval of Common Terminology Criteria (CTC) grade 1 (QTc > 0.45- 0.47 sec) or greater.
* Patients with impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

  * Left ventricular ejection fraction (LVEF) < 45% as determined by multigated acquisition (MUGA) scan or echocardiogram;
  * complete left bundle branch block;
  * obligate use of a cardiac pacemaker;
  * congenital long QT syndrome;
  * history or presence of ventricular tachyarrhythmia;
  * presence of unstable atrial fibrillation (ventricular response > 100 bpm) Patients with stable atrial fibrillation are eligible, provided they do not meet any of the other cardiac exclusion criteria;
  * clinically significant resting bradycardia (< 50 bpm);
  * right bundle branch block + left anterior hemiblock (bifascicular block);
  * angina pectoris = 3 months prior to starting study drug;
  * acute MI = 3 months prior to starting study drug; or
  * other clinically significant heart disease (e.g., congestive heart failure (CHF), uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen).
* Patients currently receiving treatment with medications known to prolong the QTc interval and/or to induce Torsades de Pointes arrhythmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of escalating doses of CYT997 when given in combination with standard carboplatin therapy (Phase Ib component) | Ongoing throughout therapy up until 30 days after last dose of CYT997
Progression-free survival at 6 months (PFS-6) utilising the dose of CYT997 identified in the Phase Ib component of this study (Phase II component) | 6 months after initiation of therapy

SECONDARY OUTCOMES:
Objective response rate (ORR) | Response is measured every second cycle of therapy
Overall survival | Baseline to study completion
Safety and tolerability | Measured continuously from study commencement through to 30 days after last dose of CYT997
Effects on pharmacodynamic markers of vascular disruption and tumour apoptosis | Measured during first cycle of therapy
Pharmacokinetic analysis of carboplatin and CYT997 in combination | Assessed during first cycle of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, MD, Study Chair — Peninsula Health; Helen Wheeler, MD, Principal Investigator — Royal North Shore Hospital; Ganessan Kichenadasse, MD, Principal Investigator — Flinders Medical Centre
Locations (4):
- Australia (4):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Gold Coast Hospital, Southport, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Monash Medical Centre, Melbourne, Victoria